CLINICAL TRIAL: NCT06823362
Title: Bioequivalence Study of Pentoxifylline 400 Mg in Sustained Release Tablets in Sustained Release Tablets in Healthy Subjects Under Fasting and Fed Conditions
Brief Title: Bioequivalence Study of Pentoxifylline 400 Mg in Healthy Subjects Under Fasting and Fed Conditions
Acronym: Pentoxifylline
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centro de Atencion e Investigacion Medica (Network)
Responsible Party: Principal Investigator, Humberto Reynales MD MSc PhD, Principal Investigator, Centro de Atencion e Investigacion Medica
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: - PENTOX-BIO-002-2022
Record Dates: First submitted 2025-01-29; First posted 2025-02-12 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Healthy; Healthy Donors
Keywords: Bioequivalence
MeSH Terms: interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1 Fasting (Active Comparator): Trental® 400 mg Fasting
  Interventions: Drug: Pentoxifylline
- 2 Fasting (Active Comparator): pentoxifylline TQ 400 mg Fasting
  Interventions: Drug: Pentoxifylline
- 1 Fed (Active Comparator): Trental® 400 mg Fed
  Interventions: Drug: Pentoxifylline
- 2 Fed (Active Comparator): pentoxifylline TQ 400 mg Fed
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Pentoxifylline — 400 mg
  Arms: 1 Fasting; 1 Fed
Drug: Pentoxifylline — 400 mg
  Arms: 2 Fasting; 2 Fed

SUMMARY:
Two bioequivalence studies of Pentoxifylline will be carried out in 40 healthy subjects, the first in a fasting condition 40 healthy subjects, the first in fasting condition and the second in postprandial condition.

postprandial condition, the two studies follow the same design: Complete crossover design, randomized, comparative of two study formulations, in single dose of 400 mg of Pentoxifylline sustained release tablets, 2 periods, with a washout time of 7 days between doses, the 7 days between doses, participation as a subject in these studies involves a risk studies involves a higher than minimal risk for subjects.

DETAILED DESCRIPTION:
To establish the main pharmacokinetic variables of the two formulations for the active formulations for the active ingredient pentoxifylline and the metabolites metabolites M1 Metabolite I (1- [5-hydroxyhexyl] -3,7- [5-hydroxyhexyl] -3,7- dimethylxanthine) and dimethylxanthine) and M5 Metabolite V (1- [3- [3-carboxypropyl] -3,7- [3-carboxypropyl] -3,7- dimethylxanthine)

ELIGIBILITY:
Inclusion Criteria:

* Men or women between 18 and 50 years of age at the time of signing the informed consent form.

informed consent. - Women who are not able to conceive, who are not pregnant or breastfeeding. (To be considered not able to conceive she must be at least 1 year postmenopausal).

postmenopausal for at least 1 year or be surgically sterile). Table 2.

* Female participants who are capable of conceiving must be using adequate contraceptive methods for the adequate contraceptive methods for the past 6 months and agree to continue using an adequate method of contraception for the adequate contraceptive method for 30 days after signing the consent form.
* Have been clinically diagnosed as healthy by the study physician.
* Subjects with clinical laboratory results within the normal range and/or fit by medical medical selection. (Table 2)
* Subjects were non-smokers for the last 3 months at the time of screening.
* Having signed the informed consent for the study.
* Body mass index between 18-30 kg/m2.
* Subject with complete contact information (cell phone and/or landline contact, address).
* Subject who has a family member or guardian with a contact telephone number.
* Subject with the availability of time to comply with the scheduled visits and activities.
* Subject who is willing to comply with the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Subject diagnosed with renal, cardiac, hepatic, immunologic, dermatologic, endocrine, gastrointestinal, neurologic or psychiatric disease, endocrine, gastrointestinal, neurological or psychiatric disease.
* Subject with diagnosis of hematological disorders, such as anemias and/or polycythemia.
* Subjects with a history of gastric surgery.
* Permanent or temporary use during the last 15 days of any type of medication. days prior to the administration of the drug, either on their own initiative or by medical prescription.

medical prescription. Except female patients who are planning regularly with the same contraceptive method.

the same contraceptive method in the last 6 months prior to the start of the present study.

the present study.

- Smoker in the last 3 months, regardless of the number of cigarettes at the time of selection.

selection.

* Consumption of xanthines from coffee, tea or chocolate during the previous 48 hours.
* Drinking alcohol in excess of 16 g 15 days prior to administration of the investigational drug.

equivalent to 1 beer or 2 glasses of wine.

* Positive test for the consumption of drugs of abuse or psychoactive substances at the time of screening or prior to administration of the (Table 2).
* Known hypersensitivity to the active substance or excipients of the test product.
* Medical history of angioedema or anaphylaxis.
* Pregnant or lactating woman.
* Subject diagnosed with human immunodeficiency virus, hepatitis B or hepatitis C positive.

hepatitis C positive.

* Having participated in clinical studies in the 4 months prior to the start of the present study.
* Having donated blood or reported blood loss of more than 500 mL in the 30 days prior to subject selection.

prior to subject selection.

* Subject has a clinically significant acute illness or temperature > 38°C within 24 hours prior to the within 24 hours prior to investigational product administration.
* Subject has a contraindication to blood collection due to bleeding or thrombotic disorders.

bleeding disorders or thrombocytopenia.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Outcome Measures | 0 to 24 hours
  Peak Plasma Concentration (Cmax)
Pharmacokinetic Outcome Measures | 0 to 24 hours
  Area under the plasma concentration versus time curve (AUC)

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Supporting Information: SAP, CSR
Time Frame: 2025 - 2035
Access Criteria: Indicate whether a proposal that describes planned analyses must be submitted or whether a data sharing agreement must be signed
URL: https://www.caimed.com/